CLINICAL TRIAL: NCT01476605
Title: The Efficacy of Prolotherapy and Platelet Rich Plasma Injections for Lateral Epicondylosis: a Pilot Study
Brief Title: Efficacy of Injection Therapy for Lateral Epicondylosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-2008-0148; G0810 (Other Grant/Funding Number: American Academy of Family Physicians-Foundation)
Record Dates: First submitted 2011-10-25; First posted 2011-11-22 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Tennis Elbow
Keywords: prolotherapy; Platelet rich plasma; tennis elbow; lateral epicondylosis
MeSH Terms: conditions — Tennis Elbow | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PrT-DMS (Active Comparator): 1.0 mL 5% morrhuate sodium + 1.5 mL 50% dextrose, 1 mL 2% lidocaine and 3.5 mL normal saline.
  Interventions: Procedure: PrT-DMS
- PrT-D (Experimental): PrT-D solution is 4 mL 50% dextrose, 3 mL normal saline, and 2 mL 2% lidocaine
  Interventions: Procedure: Dextrose prolotherapy
- Waitlist (No Intervention)
- Platelet rich plasma (Active Comparator)
  Interventions: Procedure: Platelet Rich Plasma injection

INTERVENTIONS:
Procedure: Dextrose prolotherapy — PrT-D solution is 4 mL 50% dextrose, 3 mL normal saline, and 2 mL 2% lidocaine
  Other Names: dextrose
  Arms: PrT-D
Procedure: PrT-DMS — PrT-DMS. 1.0 mL 5% morrhuate sodium + 1.5 mL 50% dextrose, 1 mL 2% lidocaine and 3.5 mL normal saline.
  Other Names: Dextrose and Morrhuate sodium PrT
  Arms: PrT-DMS
Procedure: Platelet Rich Plasma injection — Platelet rich plasma injection therapy (PRP) uses components of autologous blood to promote healing in chronically diseased joint tissues.
  Other Names: Platelet rich plasma
  Arms: Platelet rich plasma

SUMMARY:
While evidence does not identify any conventional therapy as definitive for chronic lateral epicondylosis (CLE, tennis elbow), basic science and limited pilot level trials support rigorous assessment of prolotherapy (PrT) and platelet-rich plasma (PRP) as therapy for CLE. The proposed study will conduct a pilot RCT assessing 2 PrT solutions and PRP injections commonly used in the treatment of moderate-to-severe tennis elbow using clinical, biomechanical and radiological outcomes. Data from this study will support a future confirmatory study to find an effective treatment for moderate-to-severe tennis elbow. In support of this goal, the investigators propose the following research questions.

Does PrT or PRP, compared to waitlist control:

1. improve pain- and function-dependent, CLE-specific quality of life among adults with CLE, as assessed by a validated questionnaire, the elbow-specific Patient-Rated Tennis Elbow Evaluation?
2. improve upper extremity performance among adults with CLE as assessed by a blinded assessor using elbow-specific, effort-dependent biomechanical measures of grip strength (pain-free and maximal), stiffness, effective mass and damping
3. improve the radiologic appearance of several pathologic features of CLE as evaluated using imaging studies of lateral elbow structures: ultrasound to assess a) neovascularity (color Doppler), b) hypoechogenicity (grayscale US), and c) tendon stiffness ("acousto-elastic strain gauge" technique) using standardized, 0-3 severity scales, and d) MRI to assess the overall common extensor tensor tendon disease severity using a standardized 0-3 scale?
4. provide satisfying treatment to subjects as assessed by a treatment satisfaction survey and a qualitative exit interview?

DETAILED DESCRIPTION:
CLE is a prevalent, disabling condition with significant individual and societal costs. The incidence of CLE is increasing. CLE is often refractory to care. There is limited scientific evidence to support specific therapies.

PrT and PRP show promise as effective therapy for CLE that can be performed in the primary care setting. Pilot-level RCTs of PrT and PRP for CLE have reported large absolute effect sizes. Findings from invitro and animal studies are consistent with the results of clinical trials and suggest that both therapies can improve clinical outcomes and modify disease in CLE. However, prior research is limited by lack of methodological rigor, non-validated outcome measures and lack of integrated multidisciplinary outcome measures.

Positive trends in the proposed study would suggest the effect size of PrT and PRP for CLE, and allow the calculation of a robust sample size to power an R01 study, and pilot test the use of an integrated set of outcome measures. Statistically significant positive results on clinical, biomechanical and radiological outcomes would demonstrate that PrT and PRP can treat, modify the disease of and may be a cure for CLE. Such findings would provide enormous benefits to patients through improved quality of life, reduced pain and disability, and to industry and society at large through reduced workers' injury claims and absenteeism.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years
2. diagnosis of CLE, confirmed by the PI using clinical symptoms and exam findings of tenderness over the lateral epicondyle and/or extensor tendon, and pain on 2 extensor muscle provocation tests
3. self-reported CLE-related pain for at least 6 months
4. self-reported failure of at least 2 of the 3 most common treatments for CLE (a course of NSAIDS, physical therapy or corticosteroid injections).

Exclusion Criteria:

1. current bilateral CLE
2. a corticosteroid injection in the prior 3 months or prior PrT or PRP for CLE
3. current carpal tunnel syndrome, other elbow pathology, or acute trauma of the CLE-affected upper extremity
4. self-reported history of bleeding disorders, other hematologic conditions, inflammatory arthritis, systemic nervous system disease, upper extremity surgeries or neuropathy
5. current use of opioids for pain
6. anticoagulation or immunosuppressive therapy in the prior month
7. intent to use NSAIDs or steroids
8. known allergy to dextrose, acetaminophen or lidocaine
9. MRI contraindications: non-compatible metal in the CLE-affected upper extremity or severe claustrophobia
10. unresolved litigation
11. self-reported pregnancy. Pregnant women are excluded from the study because pregnancy changes the characteristics of connective tissue including ligaments and tendons associated with CLE and, so, is an unacceptable confounder in this pilot level study. There is no report however, about dextrose, morrhuate sodium or PrT being harmful to pregnant women. Therefore we will not draw confirmatory labs to ensure that women of childbearing age are not pregnant. Rather we will accept self-report on pregnancy status at the time of consent. If a woman becomes pregnant during the study she will be dropped from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Patient rated tennis elbow evaluation (PRTEE) | 0, 16 and 32 weeks
  Validated disease specific quality of life questionnaire conducted at 0, 16 (all subjects) and 32 weeks (PrT only).The PRTEE will assess elbow related quality of life at each of the specified time points. Change in quality of life score in the study groups over time will be compared.

SECONDARY OUTCOMES:
Biomedical (grip strength), ultrasound (US) and magnetic resonance imaging (MRI) | 0 and 16 weeks
  Pain-free- and maximum-grip strengths will be using a hand dynamometer, a simple squeeze device with which the force of the subject's grip strength is recorded.US and MRI will be obtained at baseline and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David P Rabago, MD, Principal Investigator — University of Wisconsin, Department of Family Medicine; John Wilson, MD, Principal Investigator — UW Dept of Family Medicine
Locations (2):
- United States (2):
  - Northeast Family Medical Center, Madison, Wisconsin
  - University of Wisconsin General Clinical Research Center, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin Department of Family Medicine — http://www.fammed.wisc.edu